CLINICAL TRIAL: NCT03048214
Title: Effect of Infraclavicular Nerve Block Versus General Anaesthesia for Acute Postoperative Pain After Distal Radial Fracture Surgery
Brief Title: Effect of Nerve Block Versus General Anaesthesia for Distal Radial Fracture Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Wong Sau Ching Stanley, Clinical Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UW16-005
Record Dates: First submitted 2017-01-23; First posted 2017-02-09 (Estimated); Last update posted 2019-03-18 (Actual); Status verified 2019-03

CONDITIONS: Acute Pain
Keywords: Nerve block; Infraclavicular; Acute pain
MeSH Terms: conditions — Acute Pain | interventions — Anesthesia, General

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anaesthesia (Sham Comparator): Patients would receive routine general anaesthesia for their distal radial fracture surgery
  Interventions: Procedure: General anaesthesia
- Regional Anaesthesia (Experimental): Patients would receive routine infraclavicular nerve block for their distal radial fracture surgery
  Interventions: Procedure: Infraclavicular nerve block

INTERVENTIONS:
Procedure: Infraclavicular nerve block — Infraclavicular nerve block is a relatively safe and straightforward brachial plexus nerve block that can be used to provide intraoperative regional anaesthesia for upper limb surgeries from the elbow to fingers.
  Arms: Regional Anaesthesia
Procedure: General anaesthesia — Usual practice for upper limb surgeries.
  Arms: General Anaesthesia

SUMMARY:
This study aims to investigate whether infraclavicular nerve block improves acute postoperative pain after distal radial fracture surgery.

DETAILED DESCRIPTION:
A single blinded randomized control trial will be performed to compare regional anaesthesia with single shot infraclavicular nerve block versus general anaesthesia.

The primary outcome was postoperative NRS pain score (0-10) with movement at 24 hours after surgery. No suitable references for postoperative NRS pain scores at 24 hours that could be used for sample size calculation was found. Based on a previous study on RA versus GA for hand surgery, the standard deviation estimate of the treatments for sample size calculation was 2.86. To detect a difference in NRS pain score of 2.4/10 at a significance level of 0.05 and a power of 0.80, the minimum number of patients required per group was 23. A difference of 2.4 in NRS pain score was chosen because this has been shown to correspond to 'much improvement' in pain relief, which is clinically significant. To take into account for possible dropouts, 26 patients were recruited into each group.

Patients will be approached in the general ward before operation. The aims of the study and need for follow up assessment would be explained and patient will be recruited only if s/he agrees. After agreeing to join the study, patients will be randomly allocated to one of two groups: 1) General anaesthesia (GA) 2) Regional Anaesthesia with infraclavicular block (RA). Outcomes of patients in receiving general anaesthesia (GA) will be compared with patients receiving infraclavicular nerve block (RA).

Data Analysis Intention-to-treat will be used. Patients will remain in their initial designated groups for data analysis even if there is a change in surgical or anaesthetic/analgesic management, as long as they are undergoing distal radial fracture surgery not involving another operative site (eg bone graft). Patients in the RA group who required conversion to general anaesthesia due to inadequate infraclavicular block would remain in the RA group for data analysis.

Statistical methods used:

* Incidence of chronic post surgical pain: Chi-Square test
* NRS pain scores at 3 and 6 months after surgery: Mann-Whitney test to look at difference in mean pain scores between two groups
* duration of anaesthetic, analgesic and surgical procedures, time to extubation, cumulative opioid consumption, dose and frequency of rescue analgesic used, time to food intake and ambulation, time to discharge, patient satisfaction: Kruskal-Wallis test
* Acute NRS pain scores over 48 hours: Postoperative NRS pain scores were expressed in median (interquartile range) and analyzed using Mann-Whitney U test with post-hoc multiple comparisons using Bonferroni procedure
* Patient demographic data: One way ANOVA and chi-square test.
* Intraoperative vital signs, HRQOL, HADS, DASH-HKPWH: Repeated measures ANOVA (with Bonferroni correction when appropriate)
* Side effects and postoperative complications: Chi Square test
* When a significant result is obtained, t-test or Mann-Whitney test for numerical values and Chi-square test for categorical data will be applied for post hoc pairwise comparisons.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III
* Age 18-80 years old
* Scheduled for distal radial fracture surgery (ie open reduction and internal fixation)

Exclusion Criteria:

* Surgery involving more than distal radial fracture of the affected arm
* Known allergy to opioids (including the weak opioids tramadol and dihydrocodeine), local anaesthetic drugs, non-steroidal anti-inflammatory drugs (NSAIDS) including COX-2 inhibitors, paracetamol.
* History of chronic pain
* Alcohol or drug abuse
* Impaired renal function, defined as preoperative serum creatinine level over 120 µmol/L
* Patients with liver dysfunction (Plasma bilirubin over 34 mol/L, INR >/=1.7, ALT and AST over 100U/L)
* Pre-existing neurological or muscular disorders
* Psychiatric illness
* Impaired or retarded mental state
* Not self-ambulatory before operation
* Pregnancy
* Local infection
* Patient refusal

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2018-07-13 (Actual); Study Completion 2018-12-14 (Actual)

PRIMARY OUTCOMES:
Acute postoperative pain score | At postoperative day 1
  pain score would be recorded on postoperative day 1 using numeral rating scale

SECONDARY OUTCOMES:
Chronic pain score | At postoperative 3rd month
  chronic pain score would be recorded on postoperative 3rd month using numeral rating scale
Analgesic drug consumption | On discharge day
  Total analgesic drug consumption would be recorded on discharge day base on drug record from patient record

CONTACTS AND LOCATIONS:
Overall Officials: Stanley SC Wong, MBBS, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] McCartney CJ, Brull R, Chan VW, Katz J, Abbas S, Graham B, Nova H, Rawson R, Anastakis DJ, von Schroeder H. Early but no long-term benefit of regional compared with general anesthesia for ambulatory hand surgery. Anesthesiology. 2004 Aug;101(2):461-7. doi: 10.1097/00000542-200408000-00028. PMID 15277930
- [Background] Cepeda MS, Africano JM, Polo R, Alcala R, Carr DB. What decline in pain intensity is meaningful to patients with acute pain? Pain. 2003 Sep;105(1-2):151-7. doi: 10.1016/s0304-3959(03)00176-3. PMID 14499431
- [Derived] Wong SS, Chan WS, Fang C, Chan CW, Lau TW, Leung F, Cheung CW. Infraclavicular nerve block reduces postoperative pain after distal radial fracture fixation: a randomized controlled trial. BMC Anesthesiol. 2020 May 28;20(1):130. doi: 10.1186/s12871-020-01044-4. PMID 32466746